CLINICAL TRIAL: NCT01982305
Title: Simulator Versus Cadaver Training to Perform Ultrasound-guided Axillary Nerve Bocks
Brief Title: Pilot Study of a Nerve Block Simulator for the Training in Axillary Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universitaria de Ciencias de la Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acta No. 277 Aug 6, 2012
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Arm Injuries
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simulator (Experimental): One training session with the simulator.
  Interventions: Procedure: Simulator
- Cadaver (Active Comparator): One training session with a cadaver.
  Interventions: Procedure: Cadaver

INTERVENTIONS:
Procedure: Simulator — Axillary nerve anatomy lecture plus training with the simulator.
  Arms: Simulator
Procedure: Cadaver — Axillary nerve anatomy lecture plus training with the cadaver model.
  Arms: Cadaver

SUMMARY:
The purpose of this study is to determine whether an ultrasound-guided nerve block simulator is effective for the training of the axillary block technique.

DETAILED DESCRIPTION:
Ultrasound-guided nerve blocks are becoming the standard of care in patients requiring regional anesthesia. Cost-effective training is needed for the implementation of these techniques in the global anesthesia practice. Existing simulators are expensive and not available in low income countries. The investigators aimed to test an inexpensive simulator for the training in this technique.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia residents

Exclusion Criteria:

* Previous training in regional anesthesia techniques

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Time to locate axillary nerve in a cadaver | At the end of the procedure, expected average of 30 seconds

SECONDARY OUTCOMES:
Time to identify axillary nerve in a cadaver | During the procedure, expected average of 15 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Luis E Reyes, MD, Principal Investigator — Fundacion Universitaria de Ciencias de la Salud; Luis A Muñoz, MD, Principal Investigator — Fundacion Universitaria de Ciencias de la Salud